CLINICAL TRIAL: NCT07406204
Title: Comparative Clinical Efficacy of Tofacitinib Versus Methotrexate in Severe Alopecia Areata, Alopecia Totalis, and Alopecia Universalis: A Randomized Controlled Trial
Brief Title: Tofacitinib vs Methotrexate for Severe Alopecia Areata (TOFA-MTX-AA)
Acronym: TOFA-MTX-AA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hayat Abad Medical Complex, Peshawar (Other Government)
Responsible Party: Principal Investigator, Hira Rehman, PGR, Hayat Abad Medical Complex, Peshawar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMC-DERM-TOFA-MTX-AA
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Alopecia Areata; Alopecia Totalis (AT); Alopecia Universalis
Keywords: Tofacitinib; Methotrexate; Janus Kinase Inhibitor; Severe Alopecia Areata; Autoimmune Hair Loss
MeSH Terms: conditions — Alopecia Areata; Alopecia universalis | interventions — tofacitinib; Methotrexate

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to two parallel treatment arms (tofacitinib vs methotrexate) and followed for 12 weeks. Efficacy will be assessed by change in SALT score from baseline to week 12.
Masking Description: This is an open-label trial. Due to different dosing schedules and monitoring requirements for the two interventions, blinding of participants, treating clinicians, investigators, and outcome assessors will not be feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tofacitinib 10 mg Twice Daily (Experimental): Participants will receive oral tofacitinib 10 mg twice daily for 12 weeks. Clinical response will be assessed using the SALT score at baseline and at week 12. Efficacy is defined as >50% improvement in SALT score from baseline.
  Interventions: Drug: Tofacitinib
- Methotrexate 0.2-0.4 mg/kg Weekly (Active Comparator): Participants will receive oral methotrexate 0.2-0.4 mg/kg once weekly for 12 weeks with routine follow-up and laboratory monitoring for adverse effects as per institutional protocol. Clinical response will be assessed using the SALT score at baseline and at week 12. Efficacy is defined as >50% improvement in SALT score from baseline.
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Tofacitinib — Oral tofacitinib 10 mg twice daily for 12 weeks.
  Arms: Tofacitinib 10 mg Twice Daily
Drug: Methotrexate — Oral methotrexate 0.2-0.4 mg/kg once weekly for 12 weeks, with routine monitoring for adverse effects as per institutional protocol.
  Arms: Methotrexate 0.2-0.4 mg/kg Weekly

SUMMARY:
This study will compare two oral medicines-tofacitinib and methotrexate-for treating severe alopecia areata, including alopecia totalis (loss of all scalp hair) and alopecia universalis (loss of scalp and body hair). Alopecia areata is an autoimmune condition that can cause significant hair loss and emotional distress.

Adults aged 18 to 60 years with severe disease will be enrolled at the Department of Dermatology, MTI-Hayatabad Medical Complex, Peshawar, after ethical approval and written informed consent. Participants will be randomly assigned to receive either tofacitinib 10 mg twice daily or methotrexate 0.2-0.4 mg/kg once weekly for 12 weeks.

The main outcome will be improvement in hair loss measured by the Severity of Alopecia Tool (SALT) score. Treatment will be considered effective if there is more than 50% improvement in SALT score from baseline at the end of 12 weeks. Safety will be monitored during follow-up visits. The findings may help guide treatment decisions for severe alopecia areata in our local population.

DETAILED DESCRIPTION:
This is a single-center, parallel-group, randomized controlled trial to compare the clinical efficacy of oral tofacitinib versus methotrexate in adults with severe alopecia areata, including alopecia totalis and alopecia universalis, conducted at the Department of Dermatology, MTI-Hayatabad Medical Complex, Peshawar.

After approvals from the Institutional Ethical Committee and CPSP-REU and after obtaining written informed consent, eligible participants aged 18-60 years with severe alopecia areata/totalis/universalis diagnosed by a consultant dermatologist will be enrolled using consecutive non-probability sampling. Patients already receiving systemic therapy for hair regrowth, pregnant women, and patients with renal, hepatic, or pulmonary disease (based on history and clinical assessment) will be excluded.

Baseline demographic and clinical data will be recorded, and baseline disease severity will be assessed using the Severity of Alopecia Tool (SALT) score. Participants will be randomized using blocked randomization into two treatment arms:

Arm A: Oral tofacitinib 10 mg twice daily for 12 weeks.

Arm B: Oral methotrexate 0.2-0.4 mg/kg once weekly for 12 weeks, with scheduled follow-up and laboratory monitoring for potential adverse effects as per institutional protocol.

Participants will be reviewed every 4 weeks during treatment. At the end of 12 weeks, the SALT score will be reassessed. The primary endpoint is clinical efficacy defined a priori as >50% improvement in SALT score from baseline at week 12. Safety and tolerability will be assessed through clinical review and routine monitoring during follow-up visits.

Data will be analyzed using SPSS (version 23.0). Quantitative variables (e.g., age, duration of disease, baseline and post-treatment SALT scores) will be summarized as mean ± standard deviation, and categorical variables (e.g., gender, residence, efficacy) will be presented as frequency and percentage. Efficacy between groups will be compared using the chi-square test, and stratification will be performed for age group, gender, residence, and disease duration; post-stratification chi-square testing will be applied. A p-value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18-60 years.

Clinical diagnosis of severe alopecia areata, alopecia totalis, or alopecia universalis (as per protocol/operational definition), confirmed by a consultant dermatologist.

Either sex.

Able and willing to provide written informed consent.

Exclusion Criteria:

Currently receiving or recently used any systemic treatment intended for hair regrowth for alopecia areata (e.g., systemic corticosteroids, immunosuppressants, JAK inhibitors).

Pregnant women.

History or clinical evidence of renal, hepatic, or pulmonary disease.

Any condition that, in the investigator's judgment, makes participation unsafe or interferes with adherence to the study protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Change in Severity of Alopecia Tool (SALT) Score | Week 12
  SALT score ranges from 0 to 100, with higher scores indicating greater scalp hair loss. The primary outcome is the change in SALT score from baseline to week 12, compared between the tofacitinib and methotrexate groups.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this is an investigator-initiated, single-center study and data sharing is not covered in the participant consent/IRB approvals. De-identified aggregate results will be reported in publications and presentations. De-identified data may be considered for sharing in the future upon reasonable request after publication, subject to additional ethical approvals and a data use agreement.

REFERENCES:
- [Result] Abe DT, Tashima LM, Basilio FMA, Mulinari-Brenner F. Clinical experience with oral tofacitinib in a patient with alopecia areata universalis and rheumatoid arthritis. Int J Trichology. 2020;12(4):188-90.
- [Result] Asma JK, Huma AS, Urooj M. A study on the role of tofacitinib among patients treated with alopecia areata. Pak J Med Health Sc. 2022;16(12):801-3.
- [Result] Iorizzo M, Tosti A. Emerging drugs for alopecia areata: JAK inhibitors. Expert Opin Emerg Drugs. 2018;23(1):77-81.
- [Result] Cervantes J, Jimenez JJ, DelCanto GM, Tosti A. Treatment of alopecia areata with simvastatin/ezetimibe. J Investig Dermatol Symp Proc. 2018;19(1):S25-S31.
- [Result] Strazzulla LC, Avila L, Lo Sicco K, Shapiro J. an overview of the biology of platelet-rich plasma and microneedling as potential treatments for alopecia areata. J Investig Dermatol Symp Proc. 2018;19(1):S21-S24.
- [Result] Lee S, Kim BJ, Lee YB, Lee WS. Hair Regrowth outcomes of contact immunotherapy for patients with alopecia areata: a systematic review and meta-analysis. JAMA Dermatol. 2018;154(10):1145-51.
- [Result] Ro BI. Alopecia areata in Korea (1982-1994). J Dermatol. 1995;22(11):858-64.
- [Result] Melo DF, Dutra TBS, Baggieri VMAC, Tortelly VD. Intralesional betamethasone as a therapeutic option for alopecia areata. an Bras Dermatol. 2018;93(2):311-12
- [Result] Chu TW, AlJasser M, Alharbi A, Abahussein O, McElwee K, Shapiro J, et al. Benefit of different concentrations of intralesional triamcinolone acetonide in alopecia areata: an intrasubject pilot study. J Am Acad Dermatol. 2015;73(2):338-40.
- [Result] Messenger AG, McKillop J, Farrant P, McDonagh AJ, Sladden M. British Association of Dermatologists' guidelines for the management of alopecia areata 2012. Br J Dermatol. 2012;166(5):916-26.
- [Result] Rajabi F, Drake LA, Senna MM, Rezaei N. Alopecia areata: a review of disease pathogenesis. Br J Dermatol. 2018;179(5):1033-48.
- [Result] Mirzoyev SA, Schrum AG, Davis MDP, Torgerson RR. Lifetime incidence risk of alopecia areata estimated at 2.1% by Rochester Epidemiology Project, 1990-2009. J Invest Dermatol. 2014;134(4):1141-2.
- [Result] Safavi KH, Muller SA, Suman VJ, Moshell AN, Melton LJ. Incidence of alopecia areata in Olmsted County, Minnesota, 1975 through 1989. Mayo Clin Proc. 1995;70(7):628-33
- [Result] Pratt CH, King LE, Messenger AG, Christiano AM, Sundberg JP. Alopecia areata. Nat Rev Dis Primers. 2017;3:17011.
- [Result] Gilhar A, Etzioni A, Paus R. Alopecia areata. N Engl J Med. 2012;366(16):1515-5.